CLINICAL TRIAL: NCT03778528
Title: Evaluation of Ocular Lens Proteins in Cataract From Individuals With Down Syndrome
Status: Terminated | Type: Observational
Why Stopped: researcher left the institution study will not continue
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0372
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Cataract; Down Syndrome
MeSH Terms: conditions — Cataract; Down Syndrome | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cataractous tissue removed at time of cataract surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Down syndrome: Individuals with Down syndrome undergoing cataract surgery.
  Interventions: Procedure: cataract surgery
- Control: Age-matched controls undergoing cataract surgery.
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — tissue collection.

SUMMARY:
This study involves the collection ocular lens tissue from individuals with Down syndrome and age-matched controls at the time of cataract surgery.

DETAILED DESCRIPTION:
Individuals with Down syndrome have an increased rate of cataract. The reason for this increase is unclear. Normally, once cataracts become a significant impairment, an ophthalmologist will determine when cataract surgery should be performed. When this surgery is performed, cataractous tissues are cut out and discarded with medical waste. In this study, these tissue will be collected and protein analysis performed to determine what changes in different proteins are found in Down syndrome lenses as compared to normal cataractous lenses.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cataract surgery for lens extraction.

Exclusion Criteria:

* Known genetic cause other than Down syndrome causing cataract.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with Down syndrome having cataract surgery or age-matched control.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in protein composition | one week after collection of tissue
  western blot analysis of proteins from cataractous tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Age, trisomy status, protein concentration levels